CLINICAL TRIAL: NCT00539305
Title: Testosterone Supplementation in Men With MCI
Brief Title: Hormone and Information Processing Study
Acronym: HIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Monique Cherrier, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29975-A; R01AG027156 (NIH); 1R01AG027156-01A2 (NIH)
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: selective androgen receptor modulators (SARMs); hormone replacement therapy; age-associated cognitive decline; testosterone supplementation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study drug; testosterone transdermal gel (Experimental): Dose will be adjusted as needed to maintain a target total T level of 500-900 ng/dl
  Interventions: Drug: testosterone gel
- 2 (Placebo Comparator)
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: testosterone gel — 50-100mg applied topically daily for six months
  Other Names: Solvay Testosterone Gel
  Arms: Study drug; testosterone transdermal gel
Drug: placebo gel — applied topically daily for six months
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effects of testosterone (T) replacement on changes in thinking and memory, as well as mood in older men with mild cognitive impairment (MCI) and low T levels. The study will also examine whether taking testosterone has effects on biological markers related to Alzheimer's disease.

DETAILED DESCRIPTION:
Natural age related declines in testosterone (T) are associated with decreases in cognitive abilities independent of health status. Low T levels over time are associated with increased risk for developing Alzheimer's disease (AD). These findings suggest that men with low T levels are most at risk for age-related cognitive decline and AD and therefore most likely to benefit from T supplementation to prevent the development of AD or age-associated cognitive decline. The current study will assess cognition, mood, and cerebral spinal fluid (CSF) biomarker response to T supplementation in older men with mild cognitive impairment (MCI) and low T levels.

Participants will be randomized to either receive T treatment or a placebo for six months. Participants will come in for about five visits within the span of six months where they will complete cognitive & memory tests, fill out mood questionnaires, and have their blood drawn to monitor the medication level. A sample of blood will also be taken at one visit to test for apolipoprotein E (APOE), which is a genetic risk factor associated with AD. Participants will have the option to get a spinal tap in order to measure biological markers associated with Alzheimer's disease including beta-amyloid 1-40, 42, total-tau, and phosphorylated-tau-181-231. This will require an additional two visits.

ELIGIBILITY:
Inclusion Criteria:

* Male 60-90 years of age
* Diagnosis of mild cognitive impairment (MCI)
* Low testosterone level
* Primary language is English
* Availability of an informant who knows the participant well enough to answer questions
* Stable medications for the previous 3 months
* Normal complete blood count (CBC), and no clinically significant blood chemistry
* American Urological Association (AUA) symptom score less than or equal to 19
* Body Mass Index (BMI) less than 33 and stable weight in the previous year

Exclusion Criteria:

* Prior history of prostate cancer or prostate specific antigen level greater than 4.0ng/ml
* Peripheral or vascular disease
* Significant history of alcohol abuse, current alcohol abuse (more than 2 drinks per day), or other substance abuse
* History of severe head injury (with loss of consciousness greater than 30 minutes)
* Significant neurological illness, such as Parkinson's disease, seizure disorder, multiple sclerosis, major stoke
* Smokes cigarettes
* Major psychiatric illness, such as schizophrenia or bipolar disorder

Prohibited Medications:

* Anti-convulsants
* Anti-psychotics
* Sedating antihistamines
* Sedative/hypnotics
* Benzodiazepines
* Hormone or testosterone regimens
* Gonadotropin-releasing hormone (GNRH) antagonists
* Flutamide
* Anti-depressants and/or anti-cholinesterase inhibitors, but acceptable if on stable dose for 3 months or more

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Cherrier, PhD, Principal Investigator — University of Washington
Locations (1):
- VA Puget Sound Health Care Systems, Seattle, Washington, United States

REFERENCES:
- [Background] Cherrier MM, Asthana S, Plymate S, Baker L, Matsumoto AM, Peskind E, Raskind MA, Brodkin K, Bremner W, Petrova A, LaTendresse S, Craft S. Testosterone supplementation improves spatial and verbal memory in healthy older men. Neurology. 2001 Jul 10;57(1):80-8. doi: 10.1212/wnl.57.1.80. PMID 11445632
- [Background] Cherrier MM, Matsumoto AM, Amory JK, Ahmed S, Bremner W, Peskind ER, Raskind MA, Johnson M, Craft S. The role of aromatization in testosterone supplementation: effects on cognition in older men. Neurology. 2005 Jan 25;64(2):290-6. doi: 10.1212/01.WNL.0000149639.25136.CA. PMID 15668427
- [Background] Cherrier MM, Matsumoto AM, Amory JK, Asthana S, Bremner W, Peskind ER, Raskind MA, Craft S. Testosterone improves spatial memory in men with Alzheimer disease and mild cognitive impairment. Neurology. 2005 Jun 28;64(12):2063-8. doi: 10.1212/01.WNL.0000165995.98986.F1. PMID 15985573
- [Background] Cherrier MM, Matsumoto AM, Amory JK, Johnson M, Craft S, Peskind ER, Raskind MA. Characterization of verbal and spatial memory changes from moderate to supraphysiological increases in serum testosterone in healthy older men. Psychoneuroendocrinology. 2007 Jan;32(1):72-9. doi: 10.1016/j.psyneuen.2006.10.008. Epub 2006 Dec 4. PMID 17145137
- [Background] Lu PH, Masterman DA, Mulnard R, Cotman C, Miller B, Yaffe K, Reback E, Porter V, Swerdloff R, Cummings JL. Effects of testosterone on cognition and mood in male patients with mild Alzheimer disease and healthy elderly men. Arch Neurol. 2006 Feb;63(2):177-85. doi: 10.1001/archneur.63.2.nct50002. Epub 2005 Dec 12. PMID 16344336

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Dose will be adjusted as needed to maintain a target total T level of 500-900 ng/dl
  testosterone gel : 50-100mg applied topically daily for six months
- Placebo Group: Placebo gel : applied topically daily for six months
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 10 | 12
Completed | 9 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Substance Use | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (9.1) | 70.0 (7.7) | 70.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Behavioral & Mood Measure: Profile of Mood States (POMS)
Description: Values represent self evaluation of vigor-activity. The scale compares t-scores of participants to published norms (range 0-100), and higher scores indicate elevated emotion in subscale. Higher t-scores in vigor-activity subscale are considered favorable. Month 3 and Month 6 values display change from baseline.
Time Frame: Baseline, 3 and 6 months
Population: Vigor-Activity
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 9 | 10
units on a scale
  Baseline | 57.7 (2.2) | 55.5 (2.0)
  Month 3 (Change from Baseline) | -4.5 (2.8) | -0.1 (2.4)
  Month 6 (Change from Baseline) | 1.9 (2.7) | -0.5 (2.5)

2. Primary Outcome: Cognitive Changes Measured by Neuropsychological Tests: Rey Auditory Verbal Learning Test
Description: Values represent total score in Long Delay Word List Recall. Higher score indicates higher level of functioning (range 0-15). Month 3 and Month 6 indicate change from baseline.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 9 | 10
units on a scale
  Baseline | 6.2 (1.1) | 4.9 (1.0)
  Month 3 (Change from Baseline) | 2.3 (0.9) | 0.0 (0.8)
  Month 6 (Change from Baseline) | 0.9 (0.9) | 1.5 (0.8)

3. Primary Outcome: Geriatric Depression Scale (GDS)
Description: Values represent self evaluation of depression (range 0-30). Higher scores indicate a more depressed mood. Month 3 and Month 6 indicate change from baseline.
Time Frame: Baseline, Month 3, Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 9 | 10
units on a scale
  Baseline | 7.2 (1.3) | 4.1 (1.2)
  Month 3 (Change from Baseline) | 0.7 (1.5) | 2.3 (1.3)
  Month 6 (Change from Baseline) | -2.8 (1.5) | 2.7 (2.3)

4. Primary Outcome: Short-Form Health Survey (SF-36)
Description: Self assessment of Physical Functioning in Health Survey. Higher scores indicate a higher level of functioning (range 0-100). Month 3 and 6 values represent change from baseline in subscale.
Time Frame: Baseline, Month 3, Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 9 | 10
units on a scale
  Baseline | 70.7 (10.4) | 85.6 (2.3)
  Month 3 (Change from Baseline) | 15.0 (9.4) | -3.8 (6.4)
  Month 6 (Change from Baseline) | 6.4 (8.6) | -5.4 (3.5)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10) | Placebo Group (N=12)
PSA elevated above 4.0 ng/ml (General disorders) | 1 (1) | 0 (0)
Emergency room with chest pains (General disorders) | 1 (1) | 0 (0) — Pain stopped within 10-15 minutes, patient was not admitted to hospital and is following up with his personal physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No